CLINICAL TRIAL: NCT02998203
Title: Organic Diet and Children's Health - ORGANIKO LIFE+
Brief Title: Organic Diet Intervention in Primary School Children
Acronym: ORGANIKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Konstantinos Makris, Associate Professor of Environmental Health, Cyprus University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CyprusUT
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Oxidative Stress; Inflammation
Keywords: organic diet; health; pesticides; inflammation biomarkers; oxidative stress biomarkers
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional phase (No Intervention): During the conventional phase, participants are asked to maintain their usual dietary choices for 40 days.
- Organic phase (Experimental): During the organic phase, participants are asked to follow strictly the two 20-day organic dietary menus provided to them for 40 days. The organic dietary menus were prepared by a certified dietitian. The meals of the organic phase are prepared by a certified organic restaurant and are delivered to school every day except Sunday. For the meals of breakfast and afternoon snacks, children choose their preferred options for the week on the Friday of the previous week according to a list of organic food items and the products for these meals are delivered on Saturday along with the rest meals. Parents are responsible to pick-up the organic meals from school and ensure that the participating children have access to them.
  Interventions: Dietary Supplement: Organic diet

INTERVENTIONS:
Dietary Supplement: Organic diet — Full organic diet from certified organic products as obtained from certified producers and cooked by a certified organic restaurant. five meals each day delivered to students.
  Arms: Organic phase

SUMMARY:
The study aims to evaluate the hypothesized benefits of a systematic organic diet for children, over those of a conventional diet. The specific objectives of this study are to: i) Demonstrate the decreased body burden of pesticides for those children consuming an organic diet, and ii) Evaluate the effects in specific biomarkers of inflammation and oxidative stress in children systematically consuming an organic diet.

DETAILED DESCRIPTION:
A single-blinded, randomised 2 x 2 cross-over study is conducted to evaluate the effect of a 40-day organic diet compared to a 40-day conventional diet on biomarkers of exposure (pesticides metabolites) and biomarkers of effect (oxidative stress/inflammation markers) in children. The study is approved by the Cyprus National Bioethics Committee (ΕΕΒΚ/ΕΠ/2016/25) and the Cyprus Ministry of Education and Culture (7.15.06.15/2). Written informed consent for children to participate in the study is obtained from children's parents or legal guardians. Study participants are recruited from public primary schools in Limassol, Cyprus following communication with the school's headmaster. Each school that participates in the study is randomized to one of the two study arms; conventional-organic or organic-conventional. Participants' blinding is not possible since children know which diet they have at each phase. However, all documents and urine containers are coded, so that researchers are blinded to subjects' identity and group allocation.

Participants provide 6 first morning urine samples during the duration of the study; 1 baseline sample, 2 samples in the conventional phase and 3 samples in the organic phase. Anthropometric measurements (weight, height, waist circumference) are taken at the beginning and end of the study by trained researchers at the school area. A baseline questionnaire is administered to parents at the beginning of the study through a telephone interview to collect information on demographic characteristics, pesticide use at household and children's activities. A food frequency questionnaire is administered to parents at the end of the conventional phase through a telephone interview to collect information about the food habits of the children during the 40-day conventional period. A food diary is given to parents at the beginning of the study and parents use it during the organic phase, to collect information about the compliance of the children to the organic dietary menu, the children's health status and the pesticide use at home.

In order to encourage adherence to the organic diet menu, an event is organised during the organic phase of both groups, with activities for children and free sampling of organic food products.

Descriptive statistics are used to summarize the demographic characteristics for participating children. Categorical variables are described as sample size and percentages, normally-distributed continuous variables as mean±SD and non-normal continuous variables as median and interquartile range (Q1-Q3) or the appropriate transformation is conducted, such as the log transformation. For testing whether characteristics of interest are different among groups the Student's t-test are utilized for continuous normally distributed variables and the chi-square test for categorical characteristics. For continuous data that are not normally distributed, the Wilcoxon non-parametric analysis is used instead or a transformation of the data is conducted first in order to meet the normality criterion.

Linear mixed-effects models are used to account for the correlation among repeat urine samples collected from the same child and determine whether mean pesticide metabolite and biomarkers concentrations differ between the organic phase and the conventional phase.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 10-12 years, residing in Cyprus over the last five years who consume primarily (> 80%) conventional food (non-organic).

Exclusion Criteria:

* Children with chronic conditions (e.g. diabetes, asthma) or allergies in food (e.g. gluten, lactose tolerance)

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 191 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos C Makris, Study Director — Cyprus University of Technology

IPD SHARING:
Plan to Share IPD: Yes
Following the publication of the manuscript, all relevant info is made available to the public.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following the publication of the manuscript, all relevant info is made available to the public.
Access Criteria: Following the publication of the manuscript, all relevant info is made available to the public.

REFERENCES:
- [Result] Makris KC, Konstantinou C, Andrianou XD, Charisiadis P, Kyriacou A, Gribble MO, Christophi CA. A cluster-randomized crossover trial of organic diet impact on biomarkers of exposure to pesticides and biomarkers of oxidative stress/inflammation in primary school children. PLoS One. 2019 Sep 4;14(9):e0219420. doi: 10.1371/journal.pone.0219420. eCollection 2019. PMID 31483785
- [Derived] Konstantinou C, Gaengler S, Oikonomou S, Delplancke T, Charisiadis P, Makris KC. Use of metabolomics in refining the effect of an organic food intervention on biomarkers of exposure to pesticides and biomarkers of oxidative damage in primary school children in Cyprus: A cluster-randomized cross-over trial. Environ Int. 2022 Jan;158:107008. doi: 10.1016/j.envint.2021.107008. Epub 2021 Nov 30. PMID 34991267
- Available data/document: Manuscript and supplementary files — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0219420

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Groups:
- Group 1 (Organic Period First, Then Conventional Period): Schools in Group 1 began first with the organic period and continued with the conventional period.
  The organic period was organized in two 20-day cycles with differences in the menu to allow for greater variety in the meals, so that the participants' compliance to the organic treatment would be enhanced. During the organic period, participants were asked to strictly follow the two 20-day organic dietary menus provided to them for a total of 40 days.
  During the conventional period, participants were asked to maintain their usual dietary habits and choices (>80% conventional diet) for a total of maximum 40 days.
- Group 2 (Conventional Period First, Then Organic Period): Schools in Group 2 began first with the conventional period and then switched to the organic period.
  During the conventional period, participants were asked to maintain their usual dietary habits and choices (>80% conventional diet) for a total of maximum 40 days.
  The organic period was organized in two 20-day cycles with differences in the menu to allow for greater variety in the meals, so that the participants' compliance to the organic treatment would be enhanced. During the organic period, participants were asked to strictly follow the two 20-day organic dietary menus provided to them for a total of 40 days.
Period: First Period (40 Days)
Arm/Group | Group 1 (Organic Period First, Then Conventional Period) | Group 2 (Conventional Period First, Then Organic Period)
Started | 67; 3 Schools | 124; 3 Schools
Completed | 43; 3 Schools | 124; 3 Schools
Not Completed | 24; 0 Schools | 0; 0 Schools
Not completed — Withdrawal by Subject | 24 | 0
Period: Second Period (40 Days)
Arm/Group | Group 1 (Organic Period First, Then Conventional Period) | Group 2 (Conventional Period First, Then Organic Period)
Started | 43; 3 Schools | 124; 3 Schools
Completed | 43; 3 Schools | 106; 3 Schools
Not Completed | 0; 0 Schools | 18; 0 Schools
Not completed — Withdrawal by Subject | 0 | 18

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Schools in Group 1 began first with the organic period and continued with the conventional period.
  The organic period was organized in two 20-day cycles with differences in the menu to allow for greater variety in the meals, so that the participants' compliance to the organic treatment would be enhanced. During the organic period, participants were asked to strictly follow the two 20-day organic dietary menus provided to them for a total of 40 days.
  During the conventional period, participants were asked to maintain their usual dietary habits and choices (>80% conventional diet) for a total of maximum 40 days.
- Group 2: Schools in Group 2 began first with the conventional period and then switched to the organic period.
  During the conventional period, participants were asked to maintain their usual dietary habits and choices (>80% conventional diet) for a total of maximum 40 days.
  The organic period was organized in two 20-day cycles with differences in the menu to allow for greater variety in the meals, so that the participants' compliance to the organic treatment would be enhanced. During the organic period, participants were asked to strictly follow the two 20-day organic dietary menus provided to them for a total of 40 days.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 43 | 106 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.03 (0.53) | 11.21 (0.61) | 11.16 (0.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 59 | 73
  Male | 29 | 47 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Pesticide Metabolite 3-phenoxybenzoic Acid (3-PBA) Levels in Urine Between Organic and Conventional Periods*
Description: Percent change in pesticide metabolite 3-phenoxybenzoic acid (3-PBA) levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last sample of organic treatment period. A one-sample t-test was used to assess whether the percent change was different than zero.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: Last sample of the conventional period and the last sample of organic period, up to 40 days for each period
Population: The percent change was estimated only for the participants who completed the full course of the organic treatment, using the log-transformed, creatinine-adjusted biomarker levels.
Measure: Number (95% Confidence Interval); unit: % change
Units Other Than Participants: schools
Groups:
- % Change in 3-PBA Between Last Sample of Conventional Period and Last Sample of Organic Period: Percent change in 3-PBA levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last urine sample of organic treatment period. The percent change was estimated only for the participants who completed the full course of the organic treatment, using the log-transformed, creatinine-adjusted biomarker levels. A one-sample t-test was used to assess whether the percent change was different than zero.
Arm/Group | % Change in 3-PBA Between Last Sample of Conventional Period and Last Sample of Organic Period
Number analyzed (Participants) | 132
Number analyzed (schools) | 6
% change | 11.4 [5.7 to 17.2]
Statistical Analysis 1: Comparison: % Change in 3-PBA Between Last Sample of Conventional Period and Last Sample of Organic Period; A one-sample t-test was used to assess whether the percent change was different than zero; Test type: Other — One-sample t-test; p < 0.001, One-sample t-test

2. Primary Outcome: Overall Difference in Median 3-PBA Levels in Urine Between the Conventional and Organic Periods*
Description: Overall difference in median 3-PBA levels between the conventional and organic periods. The overall differences in the medians of biomarkers between the conventional and the organic phase were assessed with the non-parametric Wilcoxon rank sum test on the creatinine-adjusted concentrations pooling all conventional samples (including the baseline) and the organic samples for all participants, regardless of the duration for which they followed the organic treatment.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: 1 baseline sample, 2 samples in the conventional period (typical conventional diet) and 3 samples in the organic period, up to 40 days for each Period
Population: Three schools were randomly allocated to Group 1 (67 children) and the other three to Group 2 (124 children). In total, 24 children from Group 1 and 18 children from Group 2 who withdrew from the study 1-11 days after the beginning of the organic period and did not provide an organic period urine sample, were excluded from the data analysis.
Measure: Median (Inter-Quartile Range); unit: ng/g creatinine
Units Other Than Participants: schools
Groups:
- Median 3-PBA Levels in the Conventional Period: Median 3-PBA levels (creatinine-adjusted) in the conventional period by pooling all conventional samples (including the baseline) for all participants
- Median 3-PBA Levels in the Organic Period: Median 3-PBA levels (creatinine-adjusted) in the organic period by pooling all organic samples for all participants, regardless of the duration for which they followed the organic treatment.
Arm/Group | Median 3-PBA Levels in the Conventional Period | Median 3-PBA Levels in the Organic Period
Number analyzed (Participants) | 149 | 149
Number analyzed (schools) | 6 | 6
ng/g creatinine | 2088 [689 to 5273] | 576 [164 to 1681]
Statistical Analysis 1: Comparison: Median 3-PBA Levels in the Conventional Period vs Median 3-PBA Levels in the Organic Period; The overall differences in the medians of biomarkers between the conventional and the organic periods were assessed with the non-parametric Wilcoxon rank sum test; Test type: Other — non-parametric Wilcoxon rank sum test; p < 0.001, Wilcoxon rank sum test

3. Primary Outcome: Effect of Organic Treatment in 3-PBA Levels in Urine, Taking in Account the Repeated Measures and Duration of Organic Period
Description: A linear mixed-effect regression model was fitted for 3-PBA (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: ng/g creatinine (log-transformed)
Units Other Than Participants: schools
Groups:
- Linear Mixed-effect Model of Log-transformed Pesticide Metabolite 3-PBA: A linear mixed-effect regression model was fitted for 3-PBA (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Arm/Group | Linear Mixed-effect Model of Log-transformed Pesticide Metabolite 3-PBA
Number analyzed (Participants) | 149
Number analyzed (schools) | 6
ng/g creatinine (log-transformed) | -1.214 [-1.44 to -0.987]
Statistical Analysis 1: Comparison: Linear Mixed-effect Model of Log-transformed Pesticide Metabolite 3-PBA; Test type: Other — Linear mixed-effect regression model; p < 0.001, Mixed Models Analysis — Multiple testing was accounted for using the Benjamini-Hochberg method, considering 58 regression parameter tests of the aforementioned models. Q-value<0.05 were considered statistically significant (controlling the false discovery rate at 5%)

4. Primary Outcome: Overall Difference in Median 6-chloronicotininc Acid (6-CN) Levels in Urine Between the Conventional and Organic Periods*
Description: Overall difference in median 6-CN levels between the conventional and organic periods. The overall differences in the medians of biomarkers between the conventional and the organic phase were assessed with the non-parametric Wilcoxon rank sum test on the creatinine-adjusted concentrations pooling all conventional samples (including the baseline) and the organic samples for all participants, regardless of the duration for which they followed the organic treatment.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/g creatinine
Units Other Than Participants: schools
Groups:
- Median 6-CN Levels in the Conventional Period: Median 6-CN levels (creatinine-adjusted) in the conventional period by pooling all conventional samples (including the baseline) for all participants
- Median 6-CN Levels in the Organic Period: Median 6-CN levels (creatinine-adjusted) in the organic period by pooling all organic samples for all participants, regardless of the duration for which they followed the organic treatment.
Arm/Group | Median 6-CN Levels in the Conventional Period | Median 6-CN Levels in the Organic Period
Number analyzed (Participants) | 149 | 149
Number analyzed (schools) | 6 | 6
ng/g creatinine | 26 [6 to 180] | 20 [5 to 79]
Statistical Analysis 1: Comparison: Median 6-CN Levels in the Conventional Period vs Median 6-CN Levels in the Organic Period; [analysis description as in outcome 2, analysis 1]; Test type: Other — Wilcoxon rank sum test; p = 0.017, Wilcoxon rank sum test

5. Primary Outcome: Effect of Organic Treatment in 6-CN Levels in Urine, Taking in Account the Repeated Measures and Duration of Organic Period - Odds Ratio Calculated Based on the Fit of a Logistic Mixed-effect Model
Description: A logistic model was fitted for 6-CN (binary variable; above and below LOD) due to the high number of values below LOD. The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Units Other Than Participants: schools
Groups:
- Logistic Mixed-effect Model of Pesticide Metabolite 6-CN: A logistic model was fitted for 6-CN (binary variable; above and below LOD) due to the high number of values below LOD. The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Arm/Group | Logistic Mixed-effect Model of Pesticide Metabolite 6-CN
Number analyzed (Participants) | 149
Number analyzed (schools) | 6
Odds Ratio | 0.651 [0.463 to 0.917]
Statistical Analysis 1: Comparison: Logistic Mixed-effect Model of Pesticide Metabolite 6-CN; Test type: Other — Logistic mixed-effect model; p = 0.014, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Change in Oxidative Stress/Inflammation Biomarker 8-OHdG Levels in Urine Between Organic and Conventional Periods*
Description: Percent change in oxidative stress/inflammation biomarker 8-OHdG levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last sample of organic treatment period. A one-sample t-test was used to assess whether the percent change was different than zero.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: Last sample of the conventional period and the last sample of organic period, up to 40 days for each period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % change
Units Other Than Participants: schools
Groups:
- % Change in 8-OHdG Between Last Sample of Conventional Period and Last Sample of Organic Period: Percent change in 8-OHdG levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last urine sample of organic treatment period. The percent change was estimated only for the participants who completed the full course of the organic treatment, using the log-transformed, creatinine-adjusted biomarker levels. A one-sample t-test was used to assess whether the percent change was different than zero.
Arm/Group | % Change in 8-OHdG Between Last Sample of Conventional Period and Last Sample of Organic Period
Number analyzed (Participants) | 132
Number analyzed (schools) | 6
% change | 1.7 [-0.7 to 4]
Statistical Analysis 1: Comparison: % Change in 8-OHdG Between Last Sample of Conventional Period and Last Sample of Organic Period; A one-sample t-test was used to assess whether the percent change was different than zero; Test type: Other — One-sample t-test; p = 0.167, One-sample t-test

7. Secondary Outcome: Overall Difference in Median 8-OHdG Levels in Urine Between the Conventional and Organic Periods*
Description: Overall difference in median 8-OHdG levels between the conventional and organic periods. The overall differences in the medians of biomarkers between the conventional and the organic phase were assessed with the non-parametric Wilcoxon rank sum test on the creatinine-adjusted concentrations pooling all conventional samples (including the baseline) and the organic samples for all participants, regardless of the duration for which they followed the organic treatment.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ug/g creatinine
Units Other Than Participants: schools
Groups:
- Median 8-OHdG Levels in the Conventional Period: Median 8-OHdG levels (creatinine-adjusted) in the conventional period by pooling all conventional samples (including the baseline) for all participants
- Median 8-OHdG Levels in the Organic Period: Median 8-OHdG levels (creatinine-adjusted) in the organic period by pooling all organic samples for all participants, regardless of the duration for which they followed the organic treatment.
Arm/Group | Median 8-OHdG Levels in the Conventional Period | Median 8-OHdG Levels in the Organic Period
Number analyzed (Participants) | 149 | 149
Number analyzed (schools) | 6 | 6
ug/g creatinine | 323 [222 to 471] | 296 [202 to 447]
Statistical Analysis 1: Comparison: Median 8-OHdG Levels in the Conventional Period vs Median 8-OHdG Levels in the Organic Period; [analysis description as in outcome 2, analysis 1]; Test type: Other — Wilcoxon rank sum test; p = 0.07, Wilcoxon rank sum test

8. Secondary Outcome: Effect of Organic Treatment in 8-OHdG Levels in Urine, Taking in Account the Repeated Measures and Duration of Organic Period
Description: A linear mixed-effect regression model was fitted for 8-OHdG (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: ug/g creatinine (log-transformed)
Units Other Than Participants: schools
Groups:
- Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker 8-OHdG: A linear mixed-effect regression model was fitted for 8-OHdG (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Arm/Group | Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker 8-OHdG
Number analyzed (Participants) | 149
Number analyzed (schools) | 6
ug/g creatinine (log-transformed) | -0.119 [-0.213 to -0.024]
Statistical Analysis 1: Comparison: Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker 8-OHdG; Test type: Other — Linear mixed-effect regression model; p = 0.014, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

9. Secondary Outcome: Change in Oxidative Stress/Inflammation Biomarker 8-iso-PGF2a Levels in Urine Between Organic and Conventional Periods*
Description: Percent change in oxidative stress/inflammation biomarker 8-iso-PGF2a levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last sample of organic treatment period. A one-sample t-test was used to assess whether the percent change was different than zero.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: Last sample of the conventional period and the last sample of organic period, up to 40 days for each period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % change
Units Other Than Participants: schools
Groups:
- % Change in 8-iso-PGF2a Between Last Sample of Conventional Period and Last Sample of Organic Period: Percent change in 8-iso-PGF2a levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last urine sample of organic treatment period. The percent change was estimated only for the participants who completed the full course of the organic treatment, using the log-transformed, creatinine-adjusted biomarker levels. A one-sample t-test was used to assess whether the percent change was different than zero.
Arm/Group | % Change in 8-iso-PGF2a Between Last Sample of Conventional Period and Last Sample of Organic Period
Number analyzed (Participants) | 132
Number analyzed (schools) | 6
% change | 1.6 [0.2 to 2.9]
Statistical Analysis 1: Comparison: % Change in 8-iso-PGF2a Between Last Sample of Conventional Period and Last Sample of Organic Period; A one-sample t-test was used to assess whether the percent change was different than zero; Test type: Other — One-sample t-test; p = 0.023, One-sample t-test

10. Secondary Outcome: Overall Difference in Median 8-iso-PGF2a Levels in Urine Between the Conventional and Organic Periods*
Description: Overall difference in median 8-iso-PGF2a levels between the conventional and organic periods. The overall differences in the medians of biomarkers between the conventional and the organic phase were assessed with the non-parametric Wilcoxon rank sum test on the creatinine-adjusted concentrations pooling all conventional samples (including the baseline) and the organic samples for all participants, regardless of the duration for which they followed the organic treatment.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ug/g creatinine
Units Other Than Participants: schools
Groups:
- Median 8-iso-PGF2a Levels in the Conventional Period: Median 8-iso-PGF2a levels (creatinine-adjusted) in the conventional period by pooling all conventional samples (including the baseline) for all participants
- Median 8-iso-PGF2a Levels in the Organic Period: Median 8-iso-PGF2a levels (creatinine-adjusted) in the organic period by pooling all organic samples for all participants, regardless of the duration for which they followed the organic treatment.
Arm/Group | Median 8-iso-PGF2a Levels in the Conventional Period | Median 8-iso-PGF2a Levels in the Organic Period
Number analyzed (Participants) | 149 | 149
Number analyzed (schools) | 6 | 6
ug/g creatinine | 2964 [2112 to 3871] | 3028 [2300 to 3955]
Statistical Analysis 1: Comparison: Median 8-iso-PGF2a Levels in the Conventional Period vs Median 8-iso-PGF2a Levels in the Organic Period; [analysis description as in outcome 2, analysis 1]; Test type: Other — Wilcoxon rank sum test; p = 0.259, Wilcoxon rank sum test

11. Secondary Outcome: Effect of Organic Treatment in 8-iso-PGF2a Levels in Urine, Taking in Account the Repeated Measures and Duration of Organic Period
Description: A linear mixed-effect regression model was fitted for 8-iso-PGF2a (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: ug/g creatinine (log-transformed)
Units Other Than Participants: schools
Groups:
- Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker 8-iso-PGF2a: A linear mixed-effect regression model was fitted for 8-iso-PGF2a (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was included in the model since it met the threshold of p-value<0. 05.
Arm/Group | Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker 8-iso-PGF2a
Number analyzed (Participants) | 149
Number analyzed (schools) | 6
ug/g creatinine (log-transformed) | 0.408 [0.232 to 0.584]
Statistical Analysis 1: Comparison: Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker 8-iso-PGF2a; The interaction term for time and treatment was included in the models since it met the threshold of p-value<0. 05. Specifically, for the interaction term of time and organic treatment b=-0.016, 95% CI=[-0.023,-0.010], p-value=<0.001; Test type: Other — Linear mixed-effect regression model; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

12. Secondary Outcome: Change in Oxidative Stress/Inflammation Biomarker MDA Levels in Urine Between Organic and Conventional Periods*
Description: Percent change in oxidative stress/inflammation biomarker MDA levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last sample of organic treatment period. A one-sample t-test was used to assess whether the percent change was different than zero.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: Last sample of the conventional period and the last sample of organic period, up to 40 days for each period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % change
Units Other Than Participants: schools
Groups:
- % Change in MDA Between Last Sample of Conventional Period and Last Sample of Organic Period: Percent change in MDA levels between the last sample of the conventional treatment period (before the start of the organic treatment) and the last urine sample of organic treatment period. The percent change was estimated only for the participants who completed the full course of the organic treatment, using the log-transformed, creatinine-adjusted biomarker levels. A one-sample t-test was used to assess whether the percent change was different than zero.
Arm/Group | % Change in MDA Between Last Sample of Conventional Period and Last Sample of Organic Period
Number analyzed (Participants) | 132
Number analyzed (schools) | 6
% change | 0.1 [-1.1 to 1.2]
Statistical Analysis 1: Comparison: % Change in MDA Between Last Sample of Conventional Period and Last Sample of Organic Period; A one-sample t-test was used to assess whether the percent change was different than zero; Test type: Other — One-sample t-test; p = 0.913, One-sample t-test

13. Secondary Outcome: Overall Difference in Median MDA Levels in Urine Between the Conventional and Organic Periods*
Description: Overall difference in median MDA levels between the conventional and organic periods. The overall differences in the medians of biomarkers between the conventional and the organic phase were assessed with the non-parametric Wilcoxon rank sum test on the creatinine-adjusted concentrations pooling all conventional samples (including the baseline) and the organic samples for all participants, regardless of the duration for which they followed the organic treatment.
  *Note: This test does not take into account the repeated measures for each participant and the organic treatment duration. The results of the linear-mixed effect models are the ones considered (reported in a section below) as they take into account the repeated measures for each participant and the organic treatment duration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: umol/g creatinine
Units Other Than Participants: schools
Groups:
- Median MDA Levels in the Conventional Period: Median MDA levels (creatinine-adjusted) in the conventional period by pooling all conventional samples (including the baseline) for all participants
- Median MDA Levels in the Organic Period: Median MDA levels (creatinine-adjusted) in the organic period by pooling all organic samples for all participants, regardless of the duration for which they followed the organic treatment.
Arm/Group | Median MDA Levels in the Conventional Period | Median MDA Levels in the Organic Period
Number analyzed (Participants) | 149 | 149
Number analyzed (schools) | 6 | 6
umol/g creatinine | 858 [691 to 1016] | 846 [725 to 1029]
Statistical Analysis 1: Comparison: Median MDA Levels in the Conventional Period vs Median MDA Levels in the Organic Period; [analysis description as in outcome 2, analysis 1]; Test type: Other — Wilcoxon rank sum test; p = 0.338, Wilcoxon rank sum test

14. Secondary Outcome: Effect of Organic Treatment in MDA Levels in Urine, Taking in Account the Repeated Measures and Duration of Organic Period
Description: A linear mixed-effect regression model was fitted for MDA (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was considered and subsequently dropped if it did not meet the threshold of p-value<0. 05.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: umol/g creatinine (log-transformed)
Units Other Than Participants: schools
Groups:
- Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker MDA: A linear mixed-effect regression model was fitted for MDA (log-transformed, creatinine-adjusted). The model accounted for the duration and the effect of treatment. It included student-level (repeated measures within person) and school-level (multiple students clustered within each school) random intercepts with an unstructured covariance matrix. Continuous variables, other than time (days of treatment), were centered at the population means. The model included fixed effects for treatment condition (organic or conventional) and time (days of treatment), where time = 0 was used for the start of the treatment. The model was adjusted for the baseline value (first urine sample for all children) of the outcome to account for the background participant levels. An interaction term for time and treatment was included in the model since it met the threshold of p-value<0. 05.
Arm/Group | Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker MDA
Number analyzed (Participants) | 149
Number analyzed (schools) | 6
umol/g creatinine (log-transformed) | 0.189 [0.083 to 0.295]
Statistical Analysis 1: Comparison: Linear Mixed-effect Model of Log-transformed Oxidative Stress/Inflammation Biomarker MDA; The interaction term for time and treatment was included in the models since it met the threshold of p-value<0. 05. Specifically, for the interaction term of time and organic treatment b=-0.016, 95% CI=[-0.023,-0.010], p-value=0.01; Test type: Other — Linear mixed-effect regression model; p = 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed. Based on the study design and the inclusion/exclusion criteria no adverse events were expected and no adverse events were reported during the study period (up to 80 days).
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The reported compliance may not reflect the actual compliance of the children to the organic diet, as children could either not consume all meal portion, or families could provide them with extra organic food items.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT02998203/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT02998203/SAP_001.pdf